CLINICAL TRIAL: NCT06050603
Title: Spatiotemporally Precise Neuromodulation by Transcranial Magnetic Stimulation Guided by Multimodal Neuroimaging
Brief Title: MRI Guided Closed-loop TMS-EEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Fa-Hsuan Lin, Senior scientist, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SUN-5474
Record Dates: First submitted 2023-09-03; First posted 2023-09-22 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Normal Physiology; Amnestic Mild Cognitive Impairment
Keywords: Transcranial Magnetic Stimulation; Memory Impairments

STUDY DESIGN:
Masking Description: It is a within-subjects design, which means that all subjects will receive both individualized stimulation based on their functional results and generic stimulation based on the results of a meta-analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental_Aim1: Healthy Volunteers (Experimental): All participants will receive all conditions and the order of all conditions will be counterbalanced across participants. Statistical comparisons will be within-subjects.
  Interventions: Device: TMS
- Experimental_Aim2: Amnestic Mild Cognitive Impairment (Experimental): All participants will receive all conditions and the order of all conditions will be counterbalanced across participants. Statistical comparisons will be within-subjects.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — The target locations of TMS will be cortical regions defined by either anatomical landmarks or functional regions derived from the individual's functional and structural MRI for Aim 1. TMS target locations for Aim 2 and 3 are determined by Aim 1's results. These TMS target regions will be guided by a navigation system.
  TMS will be parametrically varied with combinations of pulse strength and frequencies based on experimental conditions. TMS strength will be referred to the resting motor threshold (rMT), which will be determined independently for each participant. TMS pulses will be delivered at fixed time instants for Aim 2 and at time instants based on the phase of oscillatory neural activity for Aim 3.

SUMMARY:
The goal of this interventional study is to develop an individualized approach using transcranial magnetic stimulation (TMS) in a high-precision manner. This approach will use TMS to modulate brain activity at multiple locations simultaneously. Functional magnetic resonance imaging (fMRI) and electroencephalograph (EEG) will record the responses and guide the stimulation. Specifically, the placement and orientation of TMS coils will be tailored to stimulate the targeted functional brain areas informed by fMRI. To maximize the interventional effect, stimulation pulses will be delivered based on EEG oscillations.

DETAILED DESCRIPTION:
Background:

Transcranial magnetic stimulation (TMS) is a non-invasive technique that uses a transient electromagnetic field over a small area of the scalp to alter neuronal activity. It has been approved by Health Canada for the treatment of major depressive disorder and obsessive-compulsive disorder. Despite its clinical prevalence, TMS has a response rate of less than 50% and high intra- and inter-subject variability. Even among healthy subjects, the probability of inducing neuro-modulatory effects can be as low as 50%.

Design:

Depending on the study's aims, participants will have to visit Sunnybrook Health Sciences Centre two or three times on separate days. Participants will be screened with a medical record review before their first visit.

In the first visit, participants will have a magnetic resonance imaging (MRI) session. During the MRI session, participants will be brought inside an MRI scanner to collect images, including structural and functional MRI scans. During structural scans, participants will be asked to stay inside the MRI while images are taken. During functional MRI scans, participants will be asked to take rests with eyes open, watching and/or listening to audiovisual stimuli, and respond to stimuli by button pressing. Before starting MRI scans, a short training on the task will be taken. An additional assessment and, if necessary, training sessions will be conducted to ensure that participants undergo imaging while being able to keep their heads sufficiently for acceptable fMRI data quality. Before entering the MRI room, participants will be asked to remove any metal or magnetic sensitive objects (e.g., jewelry, keys, credit cards) to ensure safety. Earplugs or earphones will be provided to participants to reduce the loud noise produced by the MRI scanner. During the MRI scans, participants will perform the same task as notified in the training session. Short breaks will be arranged between tasks. The entire MRI procedure will take approximately one hour. If electroencephalograph (EEG) is to be recorded during MRI scans, an additional one hour is needed for EEG preparation before the MRI scans. After MRI scans, participants may be asked to rate their feelings toward the audiovisual stimuli, cognitive states, and emotional states on a computer.

Participants will be asked to attend TMS-MRI experiments twice on separate days for aim 1. In the TMS-MRI session, participants will take TMS and MRI separately. For TMS, participants will be led to a treatment room and seated in a comfortable chair in a slightly reclined position. A research staff will place an electromagnetic coil softly against each participant's head. A TMS coil will painlessly deliver magnetic pulses stimulating nerve cells at predetermined intervals. Electrodes may be mounted on the participants' wrists and around the eyes to monitor muscle activities. The treatment protocol for each participant will be based on his/her MRI scans, EEG signals, or motor responses. This step may be helped by using a camera. During TMS, participants will hear clicking sounds generated by the TMS coil and may have touching or twitching senses over their faces. After TMS, participants will be brought to an MRI room for MRI scans as described above. A rating of the participant's feelings and task performance may be taken after MRI scans.

For aims 2 and 3, participants will be asked to attend a TMS-EEG-MRI experiment once. In the TMS-EEG-MRI session, participants will first undergo TMS and EEG together. Then, participants will undergo an MRI. For TMS-EEG, participants will be led to a treatment room and seated in a comfortable chair in a slightly reclined position. Each participant will be asked to wear an EEG cap. A device is then used to measure the EEG electrode locations over the cap. Then, conductive gel will be applied to EEG electrodes over the cap. Participants may feel skin scratching when the research staffs apply the conductive gel. Additional electrodes will be attached around the participants' eyes and wrists to monitor muscle movement. During TMS, a research staff will place an electromagnetic coil softly against the participant's head. A TMS coil will painlessly deliver magnetic pulses that stimulate nerve cells. The investigators will determine the treatment protocol based on each participant's MRI scans, EEG signals, or motor responses. This step may be helped by using a camera. During TMS, participants will hear clicking sounds generated by the TMS coil and may have touching or twitching senses over their faces. After TMS, participants will be brought to an MRI room for MRI scans as described above. A rating of the participants' feelings and task performance may be taken after MRI scans.

ELIGIBILITY:
Inclusion Criteria for Healthy participants:

* Ages between 18 and 65 years;
* Healthy with no history of neurological impairment;
* Normal or correct-to-normal vision.

Inclusion Criteria for aMCI patients:

* Age 50-80 years;
* MCI clinical criteria: (a) self- or informant-reported cognitive complaint; (b) preserved independence in functional abilities; and (c) absence of dementia;
* Objective cognitive impairment supported by the following measures of general cognitive function: (a) Mini-Mental State Exam (MMSE) 24-27 (inclusive); (b) Montreal Cognitive Assessment (MoCA) 18-26 (inclusive); or (c) Clinical Dementia Rating Scale score of 0.5;
* Normal or correct-to-normal vision.

Exclusion Criteria for all participants:

* Women who are pregnant or breastfeeding;
* History of seizure (childhood febrile seizures are acceptable and these subjects may be included in the study), history of epilepsy in self or first degree relatives, stroke, brain tumor, brain surgery, head injury, known structural brain lesion;
* Have metal in the eye or skull area, brain stimulator, surgical metal, clips in the brain, cochlear implants, mental fragments in the eye, as these make TMS unsafe;
* Have non-MRI compatible metal in the body, for example metallic (forromagnetic) implants (e.g., cardiac pacemaker, aneurysm clip);
* Subjects who are uncomfortable in small closed spaces (have claustrophobia), unable to lie comfortably supine for up to 1 hour, and would feel uncomfortable in the MRI machine;
* Participation in any other study involving non-invasive brain stimulation less than two weeks ago;
* Abnormal findings on neurological examination that we will perform.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity measured by fMRI | At baseline and immediately after treatment
  Functional connectivity during resting state and psychological tasks
Response accuracy to psychological tasks | At baseline and immediately after treatment
  accuracy, or rate of conditioned responses
Reaction times | At baseline and immediately after treatment

SECONDARY OUTCOMES:
EEG functional connectivity | At baseline and immediately after treatment
  Pearson correlation coefficients (r) between electrodes

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Hsuan Lin, PhD, Principal Investigator — Sunnybrook Research Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada